CLINICAL TRIAL: NCT05591846
Title: The Effect of Web-Based and Face-to-face Training Given to Office Workers on Health Beliefs and Physical Activity Levels Regarding Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Metin Yildiz, Nurse (Asst.Prof.Dr.), Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SakaryaU-metinyildiz-001
Record Dates: First submitted 2022-10-08; First posted 2022-10-24 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Face-to-face training; health belief model; obesity; office workers; physical activity; web-based training
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face training (Experimental): Face-to-face training group: In the study, the trainings were given face to face in a meeting room suitable for individuals. Documents were explained and animations and interviews were watched.
  Interventions: Behavioral: Face-to-face training; Behavioral: web-based training
- web-based training (Experimental): web-based training Group:In the study, trainings were given to individuals through the website established. Training videos, animations, interviews and documents have been added to the website.
  Interventions: Behavioral: Face-to-face training; Behavioral: web-based training
- Control group (No Intervention): Control group: No application has been made.

INTERVENTIONS:
Behavioral: Face-to-face training — Face-to-face training
  Arms: Face-to-face training; web-based training
Behavioral: web-based training — web-based training
  Arms: Face-to-face training; web-based training

SUMMARY:
Aim: This study was evaluated to compare the effects of web-based and face-to- face education given to office workers on health beliefs and physical activity levels towards obesity.

Material and Method: The research was conducted as a randomized controlled experimental study. The study population consisted of 768 office workers between February 2020 and April 2021, and the sample of the research consisted of 90 individuals selected from the population using the improbable random sampling method. "Descriptive Feature Form," "Obesity Health Belief Model Scale," "Physical Activity Questionnaire" were used to collect data. In the analysis of data; percentile distribution, chi-square, Fisher-Freeman-Halton Exact test, t-test in independent groups, Repeated Measures ANOVA Test, Friedman Test, One Way ANOVA test, Kruskall Wallis test, and post hoc analyzes (Bonferroni, Games Howell, Dunn) were used.

ELIGIBILITY:
Inclusion Criteria:

* Having a body mass index of 30 and above,
* Being able to use a computer
* Having a desk job (Group from civil servant to manager)
* Not have a physical disability that would prevent physical activity,
* For women, not being pregnant,
* Willingness to participate in the research.
* Having internet access

Exclusion Criteria:

* Using weight-loss drugs
* Going to a dietitian
* Being on a diet
* Exercising

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Physical activity level | To the participants; initial assessment was made; Evaluation was made at the end of the 3rd month; Evaluation was done at the end of the 6th month. A total of 6 months of evaluation was made.
  Physical activity level Measures: The International Physical Activity Questionnaire(IPAQ) was used.
  When evaluating the activities of individuals, it is accepted that each activity is done for at least 10 minutes. "MET-min/week" score is obtained by multiplying "metabolic equivalent (MET) value", "day" and "minute" for each activity level.
  The MET energy values for IPAQ are as follows:
  "Walk = 3.3 MET" "Moderate-intensity physical activity = 4.0 METs" "Vigorous physical activity = 8.0 METs" Insufficient physical activity level 0 < Total MET-min/week < 600 Low level of physical activity sufficient 600 ≤ Total MET-min/week < 3000 Physical activity level sufficient 3000 ≥ MET-min/week
Health Belief Model Scale in Obesity | To the participants; initial assessment was made; Evaluation was made at the end of the 3rd month; Evaluation was done at the end of the 6th month. A total of 6 months of evaluation was made.
  Health Belief Model Scale in Obesity Scale: Developed by Dedeli and Fadıloğlu in 2010, Health Belief Model Scale in Obesity Scale evaluates individuals' beliefs and attitudes towards weight loss. The cronbach alpha coefficient of the scale, which consists of a total of 32 items, is 0.80. The scores of the items belonging to each sub-scale of the scale are calculated by summing.Health Belief Model Scale in Obesity Scale sub dimensions: Importance of Health Perceived Sensitivity Perceived Severity Perceived Benefit Perceived Obstacle In the study, the increase in the score in the relevant sub-dimension indicates that the attitude in the relevant sub-dimension increased.
Body Mass Index | To the participants; initial assessment was made; Evaluation was made at the end of the 3rd month; Evaluation was done at the end of the 6th month. A total of 6 months of evaluation was made.
  Body Mass Index Measures: Measurements were made with scales and meters. Weight and height will be combined to report BMI in kg/m^2.
Effect on sitting times | To the participants; initial assessment was made; Evaluation was made at the end of the 3rd month; Evaluation was done at the end of the 6th month. A total of 6 months of evaluation was made.
  Effect on sitting times: How many hours do you sit in a day? created with the question.It was asked through the questionnaire.
  It shows that the situation worsens as the sitting time increases.

CONTACTS AND LOCATIONS:
Overall Officials: Metin YILDIZ, Dr., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dedeli Ö, Fadiloğlu C. Development and evaluation of the health belief model scale in obesity. TAF Prev Med Bull, 2011; 10: 533-542.
- [Derived] Yildiz M, Baysal HY. The effect of web-based and face-to-face training given to office workers on health beliefs and physical activity levels regarding obesity. Int J Nurs Pract. 2024 Jun;30(3):e13193. doi: 10.1111/ijn.13193. Epub 2023 Sep 2. PMID 37658755